CLINICAL TRIAL: NCT04116307
Title: Comparison of Clinical Efficacy of Enteroadsorbent Polymethylsiloxane vs Probiotic Lactobacillus Reuteri in the Treatment of Rotaviral Gastroenteritis in Infants and Toddlers.
Brief Title: Enteroadsorbent Polymethylsiloxane vs Probiotic Lactobacillus Reuteri in the Treatment of Rotaviral Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHID-03
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — polymethylsiloxane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polymethylsiloxane (Experimental): Polymethylsiloxane (Enterosgel) is given 3 x 10 g for the initial two days, and 3 x 5 g for the next three days.
  Interventions: Dietary Supplement: Polymethylsiloxane
- Lactobacillus reuteri (Active Comparator): Probiotic Lactobacillus reuteri (BioGaia) is given 3 x 20 drops (which means 3 x 400,000.000 CFU) per day for five days.
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Polymethylsiloxane
  Other Names: Enterosgel
  Arms: Polymethylsiloxane
Dietary Supplement: Lactobacillus reuteri
  Other Names: BioGaia
  Arms: Lactobacillus reuteri

SUMMARY:
This study evaluates a new drug, new enteroadsorbent polymethylsiloxane (Enterosgel) in the treatment of rotavirus gastroenteritis in children. Half of the participants received a new drug, polymethylsiloxane and half of the participants received standard treatment - probiotic L. reuteri (BioGaia).

DETAILED DESCRIPTION:
Polymethylsiloxane and probiotic L. reuteri both hasten symptoms of the rotavirus gastroenteritis but they do so by a different mode of action.

Polymethylsiloxane is an enteroadsorbent and it possibly acts by adsorption of viruses and doing so it prevents binding rotaviruses for enterocytes. Another mode of action can be forming a thin layer over the mucosal surfaces thus protects them from various damaging factors.

Probiotics help the healing of the intestinal mucosa presumably in few ways - by normalization of gut flora, by competition with pathogen bacteria for binding sites and nutrients and by stimulation of intestinal immune system.

ELIGIBILITY:
Inclusion Criteria:

1. age 6-36 months
2. proven rotavirus gastroenteritis
3. symptom duration less than 48 hours
4. informed consent of the parents/caregivers

Exclusion Criteria:

1. rotavirus vaccination
2. rotavirus infection in a patient's history
3. severe acute or chronic illness with possible influence on rotavirus gastroenteritis outcome

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Gastroenteritis symptoms duration. | 1-8 days.
  Duration of the loose stools, fever and vomiting.

SECONDARY OUTCOMES:
Duration of the hospitalization of any kind. | 30 days
  Duration of the classic hospitalization or duration of daily hospital attending.
Total number of loose stools. | 8 days
  The total number of loose stools are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Goran Tešović, MD, PhD, Principal Investigator — University Clinic for Infectious Diseases, Zagreb
Locations (1):
- University Clinic for Infectious Diseases, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data are available for ten years.

REFERENCES:
- [Derived] Markovinovic L, Knezovic I, Kniewald T, Stemberger Maric L, Trkulja V, Tesovic G. Enteroadsorbent Polymethylsiloxane Polyhydrate vs. Probiotic Lactobacillus reuteri DSM 17938 in the Treatment of Rotaviral Gastroenteritis in Infants and Toddlers, a Randomized Controlled Trial. Front Pediatr. 2020 Dec 21;8:553960. doi: 10.3389/fped.2020.553960. eCollection 2020. PMID 33409259